CLINICAL TRIAL: NCT05066035
Title: The Reversal of Residual Neuromuscular Blockade After Neostigmine and Half-dose Sugammadex: A Comparison With Standard Reversal of Full-dose Neostigmine
Brief Title: Residual Paralysis and Reversal With Routine Neostigmine Versus Half-dose Sugammadex and Routine Neostigmine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kartal Kosuyolu Yuksek Ihtisas Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ayse Baysal, Associate Professor of Anesthesiology and Reanimation, Kartal Kosuyolu Yuksek Ihtisas Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2013.3/12
Record Dates: First submitted 2021-09-09; First posted 2021-10-04 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Neuromuscular Blockade; Sugammadex; Neostigmine; Complication of Anesthesia; Postoperative Residual Curarization; Rocuronium
Keywords: Residual Curarization; Postoperative; Complication; Neuromuscular blockade; Neostigmine; Sugammadex; Rocuronium
MeSH Terms: conditions — Delayed Emergence from Anesthesia | interventions — Neostigmine; Sugammadex

STUDY DESIGN:
Intervention Model Description: Randomized prospective clinical trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The study protocol was masked to an outcomes assessor and the persons for this duty include an observer, a resident, or an anesthesia nurse during the anesthesia process but not to the care provider or the supervising physician.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Neostigmine (Active Comparator): The Group N (Neostigmine) (n=48), patients received standard intravenous neostigmine 0.05 mg/kg and atropine 0.02 mg/kg doses before extubation.
  A train-of-four (TOF) count of 2 in TOF Watch monitoring provides information of a shallow neuromuscular block. If at least two twitches are on the TOF watch monitor, the study investigators administer reversal medication for neuromuscular blockade in both groups. At this point, depending on randomization, a reversal agent is administered for each randomized group by an anesthesia resident or nurse who is blinded to the study protocol. The study investigators record the recovery periods between the start of administering the reversal agent to the recovery of TOF ratio < 0.9 to 0.7 and TOF ratio ≥ 0.9 if it occurs. These time periods are in minutes.
  Interventions: Drug: Neostigmine
- Neostigmine and Sugammadex (Active Comparator): In Group N+S (Neostigmine+Sugammadex) (n=50), patients received standard intravenous neostigmine 0.05 mg/kg and atropine 0.02 mg/kg doses before extubation. After a three-minute waiting period, the study investigators administered an intravenous bolus half-dose of 1 mg/kg of sugammadex after the standard reversal dose.
  A train-of-four (TOF) count of 2 in TOF Watch monitoring provides information of a shallow neuromuscular block. If at least two twitches are on the TOF watch monitor, the study investigators administer reversal medication for neuromuscular blockade in both groups. At this point, depending on randomization, a reversal agent is administered for each randomized group by an anesthesia resident or nurse who is blinded to the study protocol. The study investigators record the recovery periods between the start of administering the reversal agent to the recovery of TOF ratio < 0.9 to 0.7 and TOF ratio ≥ 0.9 if it occurs. These time periods are in minutes.
  Interventions: Drug: Sugammadex

INTERVENTIONS:
Drug: Neostigmine — The study investigators administer neostigmine at the end of operation to reverse neuromuscular blockade, and the routine dose of the intravenous neostigmine is 0.05 mg/kg and atropine 0.02 mg/kg. The dose is given in a single syringe, and later they administer this reversal medication before extubation.
  In the case of a residual block, the neostigmine group of patients receives a rescue dose of neostigmine at a dose of 0.03 mg/kg in the operating room fifteen minutes before discharge.
  Other Names: Routine full-dose reversal medication
  Arms: Neostigmine
Drug: Sugammadex — The study investigators administer the routine full-dose neostigmine reversal medication and three minutes later, they administer an intravenous bolus dose of 1 mg/kg sugammadex in a different syringe prepared earlier as a reversal agent. The anesthesia team considers using an intravenous rescue dose of 1 mg/kg sugammadex for this group of patients in the recovery room if patients do not show a complete recovery of TOF ratio equal to >0.9 in the recovery room before discharge to the ward.
  Other Names: Routine full-dose reversal medication and half-dose sugammadex
  Arms: Neostigmine and Sugammadex

SUMMARY:
Sugammadex may prevent residual neuromuscular blockade by providing rapid reversal at the end of the operation. Our goal is to compare the half-dose use of sugammadex for reversing residual blockade after administration of neostigmine and atropine to the routine use of reversal medication.

DETAILED DESCRIPTION:
Background: Postoperative residual neuromuscular block (PONB) may be observed in patients in the recovery room after surgery, and this event causes significant adverse events such as respiratory muscle weakness, decreased tidal volumes causing hypoxemia, reintubation, prolonged mechanical ventilation, and possible risk for a cardiopulmonary arrest.

Goal: The study investigators hypothesized to investigate the effects of the half-dose use of sugammadex for reversing residual blockade after administration of neostigmine and atropine and compare these results to the routine full-dose use neostigmine and atropine.

The Study Design:

The study investigators planned to perform a prospective, single-blinded, randomized trial.

The study Protocol:

The investigators enrolled patients undergoing lower abdominal tumor resection surgery under general anesthesia who fulfill our inclusion criteria.

The study is single-blinded because the anesthesia resident, anesthesia technician, and anesthesia personnel, including the data collector, were blinded to the randomization. The supervising anesthesiologist was also a data collector, and she was not blinded to the study protocol.

The randomization into two groups required the use of a computer system. The study investigators performed a random allocation sequence by the use of randomized block design codes that are generated from a computer. Afterward, the study investigators opened an opaque and sealed envelope that contained the generated codes and randomly divided patients into two groups. During this process, they made sure that all study personnel was blinded to the randomization.

The study investigators divide patients into two groups after the randomization process, and the groups are as follows: The first group of 48 patients is called Group N. In this group of patients, and we administer intravenous neostigmine 0.05 mg/kg and atropine 0.02 mg/kg in a single syringe before extubation. The second group of 50 patients is called Group N+S. In Group N+S, the study investigators administered the standard reversal medications of intravenous neostigmine 0.05 mg/kg and atropine 0.02 mg/kg. Three minutes later, the study 'investigators administered an intravenous bolus dose of 1 mg/kg sugammadex in a different syringe prepared earlier as a reversal agent.

The Study Measurement of Parameters. The patients require general anesthesia induction with an intermediate-acting neuromuscular blocking age, rocuronium, at a dose of 0.06 mg/kg intravenously.

After induction of anesthesia and before administration of rocuronium, the investigators monitored train-of-four (TOF) counts using a monitoring device of neuromuscular blockade at the patient's ulnar nerve. For this purpose, they placed two surface electrodes above the ulnar nerve near the wrist. To monitor the nerve stimuli at the adductor pollicis muscle using acceleromyography (TOF Watch SX, Schering-Plough Ireland, Dublin, Ireland). After induction of general anesthesia, the TOF Watch device provided 50-Hz tetanic stimulation for 5 seconds, and one minute after this tetanic stimulation, it offered a train-of-four (TOF) stimulation. Depending on the TOF-watch-related parameters, they decided to administer rocuronium, the neuromuscular agent, or not. At the end of the surgery, all anesthetics needed to be discontinued, including inhalational agents who were sevoflurane and nitrous oxide. Once the end-tidal concentration of sevoflurane reached a 0.4-0.6% level, the investigators administered the previously randomized reversal study drug.

For the administration of the reversal agents, there was a need for a TOF count of 2 observed in the TOF Watch device. A TOF count of 2 in TOF Watch monitoring provided information of a shallow neuromuscular block.

The Collected Parameters. They observed the clinical signs of recovery using several parameters. These parameters are level of consciousness, head-lift test, ability to sustain head lift, general muscle weakness, laryngospasm, and desaturation.

The study investigators collected the periods between the last dose of intravenous rocuronium and administering a reversal agent, administering a reversal agent to extubation, and administering a reversal agent to operating room discharge. These periods were in minutes. They also collected the recovery periods between the start of helping reversal agent to the recovery of TOF ratio < 0.9 to 0.7 and TOF ratio ≥ 0.9, which were in minutes.

They collected hemodynamical data, including; noninvasive mean arterial pressure, heart rate measurements, and peripheral oxygen saturation values before and subsequently at 2, 5, 10, and 30 minutes after administering the reversal drugs and in the recovery room.

The primary outcome was the incidence of a train-of-four (TOF) ratio less than 0.9 at tracheal extubation. The secondary outcomes were periods between the start of administering reversal agents and extubation or operating room discharge in minutes to achieve recovery of TOF ratio < 0.9 to 0.7 and TOF ratio ≥ 0.9.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria:
* 40 and 65 years of age,
* American Society of Anesthesiologists Physical Status (ASA-PS) of 3 and 4,
* Elective lower gastrointestinal tumor resection surgeries,
* Supine positioning,
* Surgery requiring use of general anesthesia and muscle relaxation,
* Use of inhalational agent of sevoflurane anesthesia,
* Surgical duration of about three to six hours.

Exclusion Criteria:

* History of known or suspected neuromuscular disease,
* History of renal or hepatic dysfunction,
* Hyperkalemia,
* Patients receiving antibiotics, anticonvulsants, or magnesium,
* History of stroke,
* History of glaucoma,
* History of pregnancy or breastfeeding,
* Suspicion of abdominal infection or sepsis,
* Suspected history of malignant hyperthermia,
* An allergy to medications used during general anesthesia

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2013-05-01 (Actual); Primary Completion 2016-10-01 (Actual); Study Completion 2016-12-30 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative residual neuromuscular blockade (rNMB) | After operation within 24 hours
  Incidence of postoperative residual neuromuscular blockade (rNMB) (defined as a train-of-four ratio, TOFR <0.9) measured 15 min after administration of the reversal agent.
Recovery time-1 | After operation within 120 minutes
  The comparison of the recovery periods between groups when the start of administering reversal agent to the recovery of TOF ratio < 0.9 to 0.7
Recovery time-2 | After operation within 120 minutes
  The comparison of the recovery periods between groups when the start of administering reversal agent to the recovery of TOF ratio < 0.7
Recovery time-3 | After operation within 24 hours
  The comparison of the recovery periods between groups when the start of administering reversal agent to the recovery of TOF ratio≥ 0.9
Muscle strength after extubation | After operation within 24 hours
  The clinical assessment of muscle strength in the operating room are as follows; awake status, The investigated parameters were; arousable with minimal stimulation, cooperativeness, responsive only to tactile stimulation, cooperativeness, and able to perform five-second head lift.

SECONDARY OUTCOMES:
Adverse events-1 | After operation within 24 hours
  Adverse events related to administration of reversal medications
Adverse events-2 | After operation within 24 hours
  Adverse events related to residual paralysis
Rescue medication neostigmine | After operation within 120 minutes
  A rescue dose of intravenous neostigmine at a dose of 0.03 mg/kg in the operating room after 15 minutes before discharge to recovery room.
Rescue medication sugammadex | After operation within 120 minutes
  A rescue dose of intravenous sugammadex at a dose of 1 mg/kg in the recovery room after 15 minutes before discharge to the ward from recovery room
Time frame-1 | After operation within 30 minutes
  The time period between the last dose of intravenous rocuronium and administering a reversal agent
Time frame-2 | After operation within 30 minutes
  The time period between administering a reversal agent to extubation
Time frame-3 | After operation within 60 minutes
  The time period between administering a reversal agent to operating room discharge
Time frame-4 | After operation within 120 minutes
  The time period between discharge from the operating room amd discharge from recovery room
Aldrete Score greater than nine in the recovery room | After operation within 120 minutes
  The criteria for patient discharge from the recovery room

OTHER OUTCOMES:
Noninvasive mean arterial pressure | During operation every 5 minutes and after operation in the recovery room every five minutes until discharge.
  Mean arterial blood pressure measurements during operation and after operation
Heart rate | During operation every 5 minutes and after operation in the recovery room every five minutes until discharge.
  Heart rate measurements during operation and after operation
Peripheral oxygen saturation | During operation every minute and after operation in the recovery room every minute until discharge.
  Peripheral oxygen saturation during operation and after operation

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Baysal, Principal Investigator — Kartal Kosuyolu High Speciality Training and Research Hospital

IPD SHARING:
Plan to Share IPD: Yes
We plan to share our data with individuals or organizations who reach us via phone, e-mail, or address.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: In a month after the release of the registration at https://register.clinicaltrials.gov.
Access Criteria: The study is under peer review at a journal, and after its publication, we are planning to share our data individually by responding to each request.

REFERENCES:
- [Background] Duvaldestin P, Kuizenga K, Saldien V, Claudius C, Servin F, Klein J, Debaene B, Heeringa M. A randomized, dose-response study of sugammadex given for the reversal of deep rocuronium- or vecuronium-induced neuromuscular blockade under sevoflurane anesthesia. Anesth Analg. 2010 Jan 1;110(1):74-82. doi: 10.1213/ANE.0b013e3181c3be3c. Epub 2009 Nov 21. PMID 19933538
- [Result] Puhringer FK, Gordon M, Demeyer I, Sparr HJ, Ingimarsson J, Klarin B, van Duijnhoven W, Heeringa M. Sugammadex rapidly reverses moderate rocuronium- or vecuronium-induced neuromuscular block during sevoflurane anaesthesia: a dose-response relationship. Br J Anaesth. 2010 Nov;105(5):610-9. doi: 10.1093/bja/aeq226. Epub 2010 Sep 28. PMID 20876699
- [Result] Aouad MT, Alfahel WS, Kaddoum RN, Siddik-Sayyid SM. Half dose sugammadex combined with neostigmine is non-inferior to full dose sugammadex for reversal of rocuronium-induced deep neuromuscular blockade: a cost-saving strategy. BMC Anesthesiol. 2017 Apr 11;17(1):57. doi: 10.1186/s12871-017-0348-9. PMID 28399799
- [Result] Schaller SJ, Fink H, Ulm K, Blobner M. Sugammadex and neostigmine dose-finding study for reversal of shallow residual neuromuscular block. Anesthesiology. 2010 Nov;113(5):1054-60. doi: 10.1097/ALN.0b013e3181f4182a. PMID 20885293
- [Result] Cheong SH, Ki S, Lee J, Lee JH, Kim MH, Hur D, Cho K, Lim SH, Lee KM, Kim YJ, Lee W. The combination of sugammadex and neostigmine can reduce the dosage of sugammadex during recovery from the moderate neuromuscular blockade. Korean J Anesthesiol. 2015 Dec;68(6):547-55. doi: 10.4097/kjae.2015.68.6.547. Epub 2015 Nov 25. PMID 26634077